CLINICAL TRIAL: NCT00591721
Title: Effectiveness of a Teleconference Delivered Fatigue Management Program for People With Multiple Sclerosis
Brief Title: Teleconference Fatigue Management for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Marcia Finlayson, PhD, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H133G070006
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Multiple Sclerosis
Keywords: energy conservation education; occupational therapy intervention; fatigue management; psychoeducation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy conservation education (Experimental): Participants received 6-70 minute group teleconference sessions with an occupational therapist facilitator. The intervention provided education, guided discussion, and peer support for learning about and applying energy conservation principles
  Interventions: Behavioral: Energy conservation education
- Wait list control (Other): Participants received 6-70 minute group teleconference sessions with an occupational therapist facilitator. The intervention provided education, guided discussion, and peer support for learning about and applying energy conservation principles.
  Interventions: Behavioral: Energy conservation education

INTERVENTIONS:
Behavioral: Energy conservation education — The intervention for this study is a group-based educational program delivered by teleconference to 4-6 individuals with MS by a licensed occupational therapist. The program involves 6 weekly sessions. Each session is 1 hour and 15 minutes in duration. Key topics addressed include: importance of rest, positive and effective communication, modification of the environment, using equipment and technology, setting priorities, and activity analysis and modification. Direct instruction, group discussion, and peer support are key elements of the program. Participants receive a manual with application activities that are completed in between sessions.

SUMMARY:
Approximately 60% of individuals with multiple sclerosis (MS) describe fatigue as their most disabling symptom. Energy conservation education involves teaching people with MS different strategies to manage fatigue and reduce its impact on daily life. Despite growing evidence of the effectiveness of face-to-face energy conservation education, not all people with MS are able to access these programs. The purpose of this project is to test the effectiveness and efficacy of a teleconference-delivered energy conservation education program for people with MS. The primary goals of the project are to reduce the impact of fatigue on participants' everyday lives, reduce fatigue severity, and improve quality of life. Secondary goals are to increase self-efficacy for managing fatigue and increase the number of energy conservation strategies used. The study will employ a randomly allocated two group time series design with a wait-list control group, which is one type of randomized control trial. A total of 181 people with MS will be recruited through direct mailing and advertising. The program will be delivered by telephone teleconference by a licensed occupational therapist. Outcome measures will be administered over the telephone by a research assistant before and after the program, at three months and at six months. We hypothesize that: (1) individuals in the immediate intervention group achieve better outcomes than individuals in the wait-list control group; (2) the program leads to significant reductions in fatigue impact and fatigue severity, and improved quality of life; and (3) improvements in the outcomes can be maintained over six months.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of MS
* 18 years of age or older
* functional English literacy (i.e., able to read course materials and carry on telephone conservations in English)
* Fatigue Severity Scale score of 4 or greater
* Residing in the state of Illinois

Exclusion Criteria:

* Short version - Blessed Orientation Memory Concentration Test - outside of normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia L Finlayson, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Finlayson M, Preissner K, Cho C, Plow M. Randomized trial of a teleconference-delivered fatigue management program for people with multiple sclerosis. Mult Scler. 2011 Sep;17(9):1130-40. doi: 10.1177/1352458511404272. Epub 2011 May 11. PMID 21561960
- [Derived] Finlayson M, Preissner K, Cho C. Outcome moderators of a fatigue management program for people with multiple sclerosis. Am J Occup Ther. 2012 Mar-Apr;66(2):187-97. doi: 10.5014/ajot.2012.003160. PMID 22394528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between November 2007 and April 2009 and involved the distribution of advertising through the MS Society and to Illinois residents participating in the NARCOMS volunteer MS patient registry.
Pre-assignment Details: 190 individuals were enrolled in the study (i.e., signed consent forms), but 9 of them did not complete baseline measures. Therefore 181 continued through the study.
Groups:
- Immediate Group: Participants assigned to this arm received the intervention (teleconference fatigue management) immediately after allocation.
- Wait List: Participants assigned to this arm waited 6 weeks after allocation to receive the intervention (teleconference fatigue management)
Period: Overall Study
Arm/Group | Immediate Group | Wait List
Started | 89 | 92
Completed | 68 | 70
Not Completed | 21 | 22
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Lost to Follow-up | 1 | 4
Not completed — Intervention not received | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Group | Wait List | Total
Number analyzed (Participants) | 89 | 92 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 83 | 165
  >=65 years | 7 | 9 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.1) | 53.5 (9.7) | 53.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 70 | 143
  Male | 16 | 22 | 38
Region of Enrollment [Number; unit: participants]
  United States | 89 | 92 | 181

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Subscale Scores of the Fatigue Impact Scale
Description: Fatigue impact was measured using the "Fatigue Impact Scale (FIS)" (Fisk et al, 1994). This 40-item scale evaluates the construct of perceived impact of fatigue on everyday life. Respondents rate each statement using a 5-point Likert-type scale ranging from 0 (no problem) to 4 (extreme problem). A total score (range from 0 to 160) and three subscale scores (physical - 10 items, score range 0 to 40; psychosocial - 20 items, score range 0 to 80; cognitive - 10 items, score range 0-40) can be produced from participants' responses. Higher scores reflect greater fatigue impact. What is reported here is the mean individual differences in the 7 week post subscale scores minus the baseline subscale scores
Time Frame: baseline, 7 weeks (immediate post-intervention)
Population: Intent-to-treat, imputation by maximum likelihood approach
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Group | Wait List
Number analyzed (Participants) | 89 | 92
units on a scale
  Average Change in Physical Subscale Scores | -3.74 (6.74) | -1.22 (6.24)
  Average Change in Cognitive Subscale Score | -4.24 (6.01) | -1.11 (6.18)
  Average Change in Psychosocial Subscale Score | -8.39 (11.66) | -2.38 (12.40)
Statistical Analysis 1: Comparison: Immediate Group vs Wait List; Hypothesis: Individuals who participate in the program will report significantly reduced fatigue impact immediately post-intervention compared to individuals allocated to the wait-list control group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Each baseline subscale score was subtracted from 7 week subscale score; t-tests assessed mean individual differences between groups; Mean Difference (Net) = -2.53, 95% CI 2-sided [-15.47 to 10.41], Standard Deviation 6.47

ADVERSE EVENTS:
Time Frame: Potential adverse events were monitored throughout the study, from baseline through to the final follow-up at 6 months post-intervention.
Description: No adverse events were observed at any point during the study, from baseline through to the final follow-up at 6 months post-intervention.
Arm/Group | Immediate Group | Wait List
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/92
Other Adverse Events (participants affected / at risk) | 0/89 | 0/92

LIMITATIONS AND CAVEATS:
Use of self-report rather than objective measures of MS disability. Only the participants were blinded to their allocation status. Co-intervention was tracked, but there is no way to know whether other interventions contributed to the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No